CLINICAL TRIAL: NCT00479908
Title: Investigation of the Time Course of the Interaction of the Hypotensive Effects of Sildenafil Citrate and Sublingual Glyceryl Trinitrate (GTN) in Men With Stable Angina Pectoris
Brief Title: Blood Pressure Interaction Between Sildenafil and Sublingual Glyceryl Trinitrate (GTN) in Men With Angina
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LREC/2003/8/35
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2007-05

CONDITIONS: Angina Pectoris
Keywords: Blood pressure; Angina; Sildenafil; Phosphodiesterase type 5; Organic nitrate; Glyceryl trinitrate; Drug interaction
MeSH Terms: conditions — Angina Pectoris | interventions — Sildenafil Citrate; Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sildenafil citrate
Drug: Glyceryl trinitrate

SUMMARY:
The purpose of the study is to determine for how long sildenafil potentiates the blood pressure reduction that occurs with glyceryl trinitrate in men with angina.

DETAILED DESCRIPTION:
By producing a mediator known as cGMP, nitric oxide (NO) potently dilates blood vessels. Nitrates, such as glyceryl trinitrate (GTN), are drugs that release NO (NO donors) and are widely used in the treatment and prevention of angina. Sildenafil is an effective treatment for male penile erectile dysfunction that inhibits the breakdown cGMP. When given alone it causes modest reductions in BP in healthy people and patients with cardiovascular disease. By their synergistic actions, co-administration of NO donors with sildenafil can result in large reductions in BP in patients with angina, a population at increased risk of developing erectile dysfunction. As a result, it is recommended that the two drugs not be co-administered within 24 hours of one another.

Previous studies have defined the effect of nitrates at 60 min after administration of sildenafil, the time of likely maximum interaction. However, emergency medicine physicians would value evidence of a balance of risks from which to make a personal clinical judgement about when they might consider giving GTN in a patient presenting with a severe episode of angina who has recently received sildenafil. Evidence on which to base such a judgement is currently not available. However, we have recently completed a study, showing that the interaction of GTN (0.4 mg spray) after sildenafil (100 mg) lasts less than 4 hours in healthy subjects. Whilst the findings would probably be similar for patients with angina, this question now needs to be investigated directly in order to ensure the generalisability of this work and address an important unresolved clinical issue.

Subjects will be asked to refrain from using short-acting nitrates for 24 hours and long acting nitrates for 72 hours before the start of the study. On the morning of each study visit subjects will take their normal medications, including anti-anginals, as soon as they wake up at home. They will also eat a light breakfast at home before coming to the research unit.

Subjects will attend 4 study visits, each separated by at least 5 days. At study visit 1 GTN will be administered 4 and 8 hours after oral sildenafil or matched placebo. At visit 2 GTN will be administered 4 and 8 hours after the alternative treatment (sildenafil or placebo). The order in which sildenafil and placebo are given will be randomised. At study visit 3 GTN will be administered 1 and 6 hours after sildenafil or placebo. Finally, at visit 4 GTN will be administered 1 and 6 hours after the alternative treatment (sildenafil or placebo). As with visits 1 and 2, the order in which sildenafil and placebo are given will be randomised.

Regular single measures of sitting and standing (after 2 min standing) BP and heart rate (HR) will be recorded at baseline and before and for 40 minutes after each GTN administration. Venous blood samples (20 mL) will be taken at baseline and immediately before and 40 min after each GTN administration for later determination of plasma concentrations of sildenafil and its active metabolite, UK-103,320.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Stable angina with one of:
* Classical history of exertional angina pectoris
* Previous diagnostic exercise test
* Angiographic evidence of CAD
* Aged 30 to 80 years
* Weight between 60 and 100 Kg

Exclusion Criteria:

* Regular treatment with long-acting nitrates or nicorandil where these cannot be withdrawn 72 hours prior to the study
* Myocardial infarction, unstable angina, stroke or transient cerebral ischaemia within 3 months
* Systolic BP > 170 mmHg or diastolic BP > 100 mmHg
* Systolic BP < 100 mmHg or diastolic BP < 60 mmHg
* Orthostatic hypotension (> 20 mmHg fall in systolic BP on standing)
* Diabetes treated with oral hypoglycaemic agents or insulin
* Any clinically significant disease other than stable angina, excepting other cardiovascular disease risk factors, e.g. smoking, hypercholesterolaemia and diet-controlled diabetes
* Taking any drug that interacts with sildenafil
* Evidence of drug abuse

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-01; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Effect of combined sildenafil and GTN on mean maximum reduction in blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: James J Oliver, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, Scotland, United Kingdom